CLINICAL TRIAL: NCT02741700
Title: STorytelling to Improve DiseasE Outcomes in GoUT: The STRIDE-GO Study
Brief Title: SToRytelling to Improve DiseasE Outcomes in GOut: The STRIDE-GO2 Study
Acronym: STRIDE-GO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 13-314
Record Dates: First submitted 2016-03-21; First posted 2016-04-18 (Estimated); Results first posted 2022-02-23 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Gout; Low Medication Adherence; Health Related Quality of Life
Keywords: Adherence; Disparities; Patient Outcomes
MeSH Terms: conditions — Gout

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gout storytelling video (Experimental): Participants view culturally relevant patient narrated storytelling in African-American Veterans' own voices about their experience with gout and its treatment and a patient narrated slide show of gout and its treatment.
  Interventions: Behavioral: Gout Storytelling Video Intervention
- Video about management of another chronic condition (Active Comparator): Participants view a patient narrated slide show of roughly the same duration as the experimental arm, summarizing the management of stress, a non-gout chronic condition.
  Interventions: Behavioral: Gout Storytelling Video Intervention

INTERVENTIONS:
Behavioral: Gout Storytelling Video Intervention — The investigators developed a storytelling intervention for African-Americans with gout, to address barriers to optimal gout management and provide cues for better disease management, which were narrated by several Veterans with gout. One of the veterans also presented a PowerPoint on gout and its management. The intervention was shown to the participants on a touchscreen computer or the desktop screen at the baseline study visit. Subsequently, they were provided with DVD with similar intervention to watch at home.

SUMMARY:
The objective is to test the efficacy of a patient-centered, culturally relevant narrative intervention, or "storytelling," based on the solid conceptual foundation of the narrative communication theory and the constructs of the Health Belief Model (HBM) to improve medication adherence and outcomes in chronic diseases among African-Americans (AA), using gout as an example. Gout is a chronic disease associated with chronic symptoms and disability interrupted by intermittent acute flares, similar to Chronic Obstructive Pulmonary Disease (COPD) and Congestive Heart Failure (CHF) that leads to joint destruction if not treated appropriately. Due to the intermittently symptomatic nature of chronic conditions, patients often don't perceive disease severity and susceptibility to disease complications, and, therefore, may not balance the barriers and benefits to medication adherence. Storytelling in the patients' own voices has the power to directly and more effectively confront a patient's barriers to medication adherence, reinforce the benefits and provide useful cues to action. Storytelling promotes patient engagement when the patient identifies with the storyteller and can lead to a patient's recognition of the need to treat the condition and improve health outcomes, as shown by a meaningful improvement in blood pressure in a recent clinical trial in AAs with hypertension. The success of this project, combined with other published data, will represent a major step toward demonstrating the effectiveness of storytelling to improve medication adherence in chronic diseases and will address two VA research priority areas, i.e., health care disparities and health care delivery.

DETAILED DESCRIPTION:
The investigators will conduct a 12-month, multicenter, randomized controlled trial among 250 African-American Veterans with gout with a ULT medication possession ratio of <80% at Birmingham, St. Louis, and Philadelphia VA clinics. The investigators will compare the efficacy of the storytelling intervention to usual care in improving Urate Lowering Therapy (ULT) adherence, assessed with MEMSCaps (electronic monitoring) at 6-months (primary outcome); reducing gout flares needing treatment, improving patient satisfaction, improving the ability to achieve target serum urate <6 mg/dl and improving self-reported ULT adherence at 6-months (secondary outcomes). The investigators will assess these outcomes at 12-months as evidence for the sustenance of the effect of the intervention.

Alignment with VA mission and priorities: This study serves the VA's mission of improving the health of Veterans and addresses two priority areas, 1) decreasing health care disparities and 2) improving health care delivery using a low-cost, technology-based solution to poor medication adherence. Study results will lead to a ready-to-implement low-cost patient-centered intervention for AA Veterans with gout to improve medication adherence and patient outcomes. This study will provide proof of the efficacy of "storytelling" for improving medication adherence in chronic symptomatic diseases. The "storytelling" intervention can be easily adapted for similar chronic symptomatic conditions such as COPD and CHF.

ELIGIBILITY:
Inclusion Criteria:

* African American Veteran Patients with Gout currently on urate-lowering therapy (ULT; most commonly allopurinol) with either low ULT adherence, defined as an average medication possession ration (MPR) <0.80 or MPR >=0.80

Exclusion Criteria:

* participants who use pill-box for ULT medication use
* participants who Opt-out for the research will not be contacted

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jasvinder A Singh, MD MPH, Principal Investigator — Birmingham VA Medical Center, Birmingham, AL
Locations (3):
- United States (3):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Data are owned by the VA. only with the conditions and approvals from appropriate VA authorities, we are willing to share de-identified data with requesters.

REFERENCES:
- [Derived] Singh JA. SToRytelliing to Improve Disease outcomes in Gout (STRIDE-GO) in African American veterans with gout: a trial study protocol. Trials. 2021 Dec 4;22(1):879. doi: 10.1186/s13063-021-05847-9. PMID 34863255
- [Derived] Singh JA, Joseph A, Baker J, Richman JS, Shaneyfelt T, Saag KG, Eisen S. SToRytelling to Improve Disease outcomes in Gout (STRIDE-GO): a multicenter, randomized controlled trial in African American veterans with gout. BMC Med. 2021 Nov 9;19(1):265. doi: 10.1186/s12916-021-02135-w. PMID 34749717

RESULTS

PARTICIPANT FLOW:
Groups:
- Gout Storytelling Video: Patients view a culturally relevant patient storytelling in African-American Veterans' own voices about gout and its treatment.
  Improvement of Medication Adherence: The investigators have developed a storytelling intervention for African-Americans with gout, to address barriers to optimal gout management and provide cues for better disease management. The objective of this study is to assess the efficacy of a novel storytelling intervention in Veteran's own voices to improve medication adherence and patient outcomes in African-American Veterans with gout.
- Video About Management of Another Chronic Condition: Patient narrated slide show of roughly the same duration as the experimental arm, summarizing management of a non-gout condition.
  Improvement of Medication Adherence: The investigators have developed a storytelling intervention for African-Americans with gout, to address barriers to optimal gout management and provide cues for better disease management. The objective of this study is to assess the efficacy of a novel storytelling intervention in Veteran's own voices to improve medication adherence and patient outcomes in African-American Veterans with gout.
Period: Overall Study
Arm/Group | Gout Storytelling Video | Video About Management of Another Chronic Condition
Started | 152 | 154
Completed | 126 | 135
Not Completed | 26 | 19
Not completed — Lost to Follow-up | 17 | 8
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Physician Decision | 3 | 0
Not completed — Moved out of State | 0 | 1
Not completed — Death | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gout Storytelling Video | Video About Management of Another Chronic Condition | Total
Number analyzed (Participants) | 152 | 154 | 306
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (8.3) | 65 (8.0) | 64 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 152 | 154 | 306
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 152 | 154 | 306
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 152 | 154 | 306

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence
Description: ULT adherence, directly measured by using MEMS (Medication Event Monitoring System) Caps at 3, 6, and 9 months (assess intervention's effect) and 12 months (assess the durability of effect)
Time Frame: 3, 6, 9, and 12 months
Measure: Mean (95% Confidence Interval); unit: percentage of days ULT was taken
Arm/Group | Gout Storytelling Video | Video About Management of Another Chronic Condition
Number analyzed (Participants) | 152 | 154
percentage of days ULT was taken
  MEMSCap™ ULT MPR at 3-months | 72.61 [67.88 to 77.35] | 70.12 [65.49 to 74.75]
  MEMSCap™ ULT MPR at 6-months | 68.52 [63.40 to 73.64] | 69.33 [64.36 to 74.30]
  MEMSCap™ ULT MPR at 9-months | 65.85 [60.14 to 71.55] | 67.32 [61.84 to 72.80]
  MEMSCap™ ULT MPR at 12-months | 60.54 [54.29 to 66.79] | 63.82 [57.83 to 69.82]

2. Secondary Outcome: Gout Flares
Description: Participant-reported total number of gout flares in the last 1 month
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Self-reported gout flares in 1 month
Arm/Group | Gout Storytelling Video | Video About Management of Another Chronic Condition
Number analyzed (Participants) | 152 | 154
Self-reported gout flares in 1 month | 0.74 [0.45 to 1.02] | 0.99 [0.72 to 1.26]

3. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction with medication on the patient questionnaire (SATMED composite score), range 0-100. The SATMED-Q contains 17 items, each scored on a 5-point Likert scale. The total composite score ranges between 0 and 68. The score was converted to a percentage as recommended (=(raw score*100)/68); higher score = more satisfaction with medication.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Gout Storytelling Video | Video About Management of Another Chronic Condition
Number analyzed (Participants) | 152 | 154
units on a scale | 62.16 [57.09 to 67.23] | 67.43 [62.39 to 72.47]

4. Secondary Outcome: Target Serum Urate
Description: Serum urate with absolute value in mg/dl, as indirect measures of better ULT adherence and important gout outcomes
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Gout Storytelling Video | Video About Management of Another Chronic Condition
Number analyzed (Participants) | 152 | 154
mg/dL | 5.94 [5.61 to 6.27] | 5.72 [5.41 to 6.04]

ADVERSE EVENTS:
Time Frame: 1-year
Arm/Group | Gout Storytelling Video | Video About Management of Another Chronic Condition
All-Cause Mortality (participants affected / at risk) | 4/152 | 5/154
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/154
Other Adverse Events (participants affected / at risk) | 9/152 | 5/154
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gout Storytelling Video (N=152) | Video About Management of Another Chronic Condition (N=154)
Medication side effect on SATMED-Q side effect (Product Issues) | 9 (9) | 5 (5) — Medication side effect on SATMED-Q side effect question- side effects not specified

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT02741700/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT02741700/ICF_001.pdf